CLINICAL TRIAL: NCT02927912
Title: Multi-institution Phase II Trial of Intraoperative Electron Beam Radiotherapy Boost at the Time of Breast Conserving Surgery With Oncoplastic Reconstruction in Women With Early-Stage Breast Cancer
Brief Title: Intraoperative Electron Beam Radiotherapy Boost in Treating Patients With Stage I-II Breast Cancer Undergoing Surgery With Reconstruction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sachin Jhawar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-16106; NCI-2016-01294 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Radiotherapy; Radiation; Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (IOERT boost) (Experimental): Patients undergo standard of care lumpectomy and then undergo 1 fraction of IOERT boost to the lumpectomy cavity. Patients then undergo standard of care oncoplastic reconstruction and whole breast radiation therapy.
  Interventions: Radiation: Electron Beam Therapy; Procedure: Lumpectomy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Reconstructive Surgery

INTERVENTIONS:
Radiation: Electron Beam Therapy — Undergo IOERT boost
  Other Names: photon beam radiation therapy
Procedure: Lumpectomy — Undergo lumpectomy
  Other Names: Lumpectomy of Breast; Partial Mastectomy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo whole breast radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Reconstructive Surgery — Undergo oncoplastic reconstruction
  Other Names: Reconstruction

SUMMARY:
This phase II trial studies the side effects of intraoperative electron beam radiotherapy boost and to see how well it works in treating patients with stage I-II breast cancer undergoing surgery with reconstruction. Giving a single dose of electron beam radiation to the tumor cavity during the breast surgery before reconstruction may be a better way to kill tumor cells and shrink tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of grade 3 breast fibrosis at 1 year in women undergoing lumpectomy with oncoplastic reconstruction and immediate intraoperative electron radiotherapy boost followed by adjuvant whole breast radiotherapy.

SECONDARY OBJECTIVES:

I. To determine the rate of 5 year ipsilateral breast tumor recurrence rate. II. To determine the change in self-reported cosmesis using the Breast Cancer Treatment Outcome Scale (BCTOS) questionnaire.

III. To evaluate physician-reported cosmetic outcomes using the 4-point Harvard Cosmesis Scale and digital photographs.

OUTLINE:

Patients undergo standard of care lumpectomy and then undergo 1 fraction of intraoperative electron beam radiation therapy (IOERT) boost to the lumpectomy cavity. Patients then undergo standard of care oncoplastic reconstruction and whole breast radiation therapy.

After completion of study treatment, patients are followed up at 1 month, 6 months, 1 year, and every year thereafter for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of breast cancer
* Clinical node negative stage I (T1N0) or stage II (T2N0) breast cancer

  * Preoperative ultrasound of the axilla with biopsy of suspicious nodes is recommended as clinically indicated per the discretion of the treating physician
* Appropriate stage for protocol entry including no clinical evidence for distant metastases based upon the following minimum diagnostic workup
* History/physical examination, documentation of weight and Zubrod performance status 0-2 within 28 days prior to study entry
* Right and left mammography within 90 days of diagnostic biopsy establishing diagnosis
* Absolute neutrophil count > 1800 cells/cubic mm
* Platelets >= 75,000 cells/cubic mm
* Hemoglobin >= 8 g/dL
* Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days of study entry
* Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during radiation therapy
* Patients must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Clinical T4, N2 or N3, M1 pathologic stages III or IV breast cancer
* Prior invasive non-breast malignancy (except non-melanoma skin cancer, carcinoma in situ of the cervix) unless disease free for a minimum of 3 yrs prior to study entry
* Prior invasive or in-situ carcinoma of the breast (prior lobular breast carcinoma in situ [LCIS] is eligible)
* Two or more cancers not resectable through a single lumpectomy incision
* Bilateral breast cancer
* Ductal breast carcinoma in situ (DCIS) only
* Non-epithelial breast malignancies such as sarcoma/lymphoma
* Male breast cancer
* Paget's disease of the nipple
* Prior radiotherapy to the breast or prior radiation to the region of the ipsilateral breast that would result in overlap of radiation fields
* Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
* Active systemic lupus, erythematosus, or any history of scleroderma, dermatomyositis with active rash
* Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events in the first 30 patients enrolled as graded by the National Cancer Institute Common Toxicity Criteria version 4.0 | Up to 30 days after surgery and IOERT boost
  If 4 or more complications in the first 10 patients, 7 or more out of the first 20 patients or 9 or more out of 30 patients are observed, then the study will be deemed not safe to continue. Summary statistics will be used to report all complications.
Rate of grade 3 fibrosis using the Late Effects Normal Tissue Task Force-Subjective, Objective, Management, Analytic scales | At 1 year from the end of therapy
  The proportion of patients with an overall response rate of grade 3 fibrosis at 1 year from the end of therapy along with the exact binomial confidence interval for the rate will be calculated.

SECONDARY OUTCOMES:
Change in self-reported cosmesis using the BCTOS | Baseline up to 3 years
  The mean and standard deviation of the self-reported cosmesis using the BCTOS cosmesis scale will be summarized over time. The change over time using a repeated measures model or non-parametric methods, if appropriate, will be examined.
Physician reported cosmesis using the Harvard Breast Cosmesis scale and digital photographs | Up to 3 years after completion of radiation therapy
  physician-reported cosmetic outcomes using the 4-point Harvard Cosmesis Scale and digital photographs
Quality of life assessed by Breast Cancer Treatment Outcome Scale | Up to 3 years after completion of radiation therapy
  determine the rate of surgical complications necessitating hospital readmission or return to the operating room within 30 days of surgery + IOERT
Rate of ipsilateral breast tumor recurrence | At 5 years
  The exact binomial confidence interval for the rate will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bazan, MD, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (5):
- United States (4):
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
- Centre Hospitalier de I'Universite de Montreal, Québec, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu